CLINICAL TRIAL: NCT00901407
Title: Lamotrigine as an Antidepressant Augmentation Agent in Treatment Refractory Unipolar Depression
Brief Title: Lamotrigine Augmentation in Resistant Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Louisiana State University Health Sciences Center in New Orleans (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: James G. Barbee, IV, MD, LSUHSC
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LMC-R93
Record Dates: First submitted 2009-05-11; First posted 2009-05-13 (Estimated); Last update posted 2009-05-13 (Estimated); Status verified 2009-05

CONDITIONS: Unipolar Depression
Keywords: augmentation; depression; resistance
MeSH Terms: conditions — Depressive Disorder; Depression | interventions — Lamotrigine; Paroxetine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): lamotrigine
  Interventions: Drug: lamotrigine; Drug: paroxetine
- 2 (Placebo Comparator): placebo
  Interventions: Drug: placebo; Drug: paroxetine

INTERVENTIONS:
Drug: lamotrigine — lamotrigine augmentation 25 to 100 mg tablets, 25 to 200 mg bid,10 weeks
  Other Names: Lamictal
  Arms: 1
Drug: placebo — placebo: 1-2 tablets bid; 10 weeks
  Arms: 2
Drug: paroxetine — open label paroxetine 10 to 50 mg, at bedtime for 18 weeks (8 weeks prior to randomization and 10 weeks after)
  Other Names: paxil

SUMMARY:
This study is intended to evaluate the efficacy and safety of lamotrigine as an antidepressant augmentation agent in a sample of individuals with major depression and a history of both prior non-response and prospective failure to respond to at least one adequate trial of an antidepressant (for a total of two failed trials).

DETAILED DESCRIPTION:
The study will consist of four phases: screening, open-label, double-blind and discontinuation phases. After screening to ensure that subjects meet the study criteria, individuals will enter an open-label (flexible-dose) trial of paroxetine-CR given in dosages up to 62.5 mg for a period of eight weeks. Paroxetine may be substituted for paroxetine-CR in dosages up to 50 mg. Subjects may be switched from paroxetine-CR to the bioequivalent dose of paroxetine due to drug supply disruption but should not be switched back to paroxetine-CR. Subjects are not allowed to switch from paroxetine to paroxetine-CR. Subjects who start on paroxetine at the first visit must remain on paroxetine for the duration of the study. At the discretion of the investigator, additional monitoring or interim visits may be needed for subjects who require a switch from paroxetine-CR to paroxetine. Those individuals who fail to respond adequately will then continue into the second phase (double-blind portion) of the study, in which participants will continue on either paroxetine-CR or paroxetine, and will be randomized to either placebo or lamotrigine in a flexible-dose design up to 400mg for a 10-week period. Subjects will remain on the same dose of paroxetine-CR or paroxetine that they were taking at the final visit in the first phase of the study (Visit 5/Week 8). The study medications will be discontinued following the final study visit (Visit 11/Week 18 or the early termination visit). Paroxetine-CR or paroxetine may be continued in the dosages used during the study after completion of the protocol if, in the judgment of the investigator, the subject has shown a partial response to treatment with the drug. The lamotrigine (or placebo) dose will be decreased by half for one week and then discontinued. Subjects will return two weeks post-study and four weeks post study for follow up visits consisting of safety evaluations. In addition, a MADRS and CGI should be performed at the two-week post study follow up visit. The visit at four weeks post study may be omitted if the 3rd and 4th week of taper are not needed. The decision to restart lamotrigine at that time would also be up to the investigator, but the dosage of lamotrigine would have to be titrated in the first month per the manufacturer's clinical trial program. This is necessary since all subjects will be discontinuing from the drug following Visit 11/Week 18 or the early termination visit in order to maintain the blind at the conclusion of each subject's participation in the study. Subjects who are discontinued from paroxetine-CR at dosages of 25 mg/day or higher should undergo a gradual dose reduction of 12.5 mg per week rather than abrupt cessation. Subjects who are discontinued from paroxetine at dosages of 20 mg/day or higher should undergo a gradual dose reduction of 10 mg per week rather than abrupt cessation.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects, age 18-65
2. A current primary diagnosis of unipolar major depression based on certain criteria
3. Have a score of > 18 on the 17-item Hamilton Depression scale
4. A history of prior failure of at least one adequate trial of an FDA-approved antidepressant. The antidepressant failure must have occurred within the current episode of major depression
5. Females of childbearing potential will be allowed as long as they are taking adequate contraceptive precautions

Exclusion Criteria:

1. A primary Axis I diagnosis other than primary unipolar major depression
2. A history suggestive of hypomania or mania during the current episode or during the person's lifetime
3. A history of psychosis, dementia, organic affective disorders or alcohol and/or substance abuse in the previous six months

   * Individuals with a current or past diagnosis of schizoid, schizotypal, borderline or antisocial or any other current or past severe personality disorder
   * Individuals with a current or past diagnosis of schizophrenia or schizoaffective disorder
4. A history of failure to respond to electroconvulsive therapy during the current or any prior lifetime episode of major depression
5. A history of failure of a prior adequate trial of paroxetine or paroxetine-CR for the treatment of Major Depression
6. Significant, coexisting medical conditions that might make it unsafe to take either of the study medications, or in which any average reasonable clinician would assume that the medical condition may, in fact, be exacerbating the current episode of depression or impede the person's ability to recover fully from their depressive illness
7. Presence of significant medical abnormalities on baseline laboratory values or physical examination, including vital signs

   * Individuals with any significant abnormalities of thyroid function
   * Subjects on thyroid supplementation must have been on a stable dose for six months prior to the screening visit
8. Individuals who will require concomitant psychotropic medications, including benzodiazepines

   * Subjects with severe insomnia will be allowed to take a maximum of 10 mg of zolpidem on two nights weekly at the investigator's discretion.
   * Zolpidem may not be taken on the night before the study visit.
   * Each dose of zolpidem should be listed on the concurrent medication case report form
9. Medications likely to cause significant effects on mood and anxiety are also excluded
10. Individuals with a positive urine drug screen for drugs of abuse at the screening visit
11. Use during the time of the study of any medications known to affect the metabolism of lamotrigine

    * Individuals on valproate and carbamazepine will be specifically excluded
    * Investigators should be aware that oral contraceptives have been reported to lower the levels of lamotrigine, but any change in dosing is left to the judgment of the investigator
12. Subjects who have taken other psychoactive drugs within certain time frames of the screening visit
13. The presence of significant risk of suicide
14. Pregnant females or those who are breastfeeding infants
15. A history of hypersensitivity or intolerance to either of the study medications, lamotrigine or paroxetine or paroxetine-CR
16. Subjects initiating or terminating psychotherapy within 12 weeks of the screening visit
17. Individuals who are currently on disability for a psychiatric disorder, or who are in any other way likely to experience considerable secondary gain from the persistence of their psychiatric illness, such as pending legal litigation of any type
18. Individuals who in the opinion of the investigator would not be able to understand or comply with the study requirements

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2003-12; Primary Completion 2006-07 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
MADRS score | weeks 0 (randomization); 8, 9, 10, 12, 14, 16, 18, and 20

SECONDARY OUTCOMES:
Ham-D score | weeks 0 (randomization); 2, 4, 6, 8, 9, 10, 12, 14, 16, and 18
CGI-S and CGI-I | weeks 0 (randomization); 8, 9, 10, 12, 14, 16, 18 and 20

CONTACTS AND LOCATIONS:
Overall Officials: James G. Barbee, MD, Principal Investigator — Louisiana State University Health Sciences Center in New Orleans
Locations (1):
- LSUHSC- New Orleans, New Orleans, Louisiana, United States

REFERENCES:
- [Result] Barbee, J.G., Jamhour, N,J., Stewart, J.W., Shelton, R.C., Reimherr, F.W., Thompson, P.M., Conrad, E.J. &Thompson, T.R. (2007, May). Lamotrigine as an antidepressant augmentation in treatment refractory unipolar depression. Poster session presented at the annual meeting of the American Psychiatric Association, San Diego, CA.
- [Result] Barbee, J.G., Jamhour, N,J. & Conrad, E.J. (2007, June). Predictors of response to lamotrigine augmentation in treatment refractory unipolar depression. Poster session presented at the annual meeting of the New Clinical Drug Evaluation Unit, Boca Raton, FL.
- [Derived] Barbee JG, Thompson TR, Jamhour NJ, Stewart JW, Conrad EJ, Reimherr FW, Thompson PM, Shelton RC. A double-blind placebo-controlled trial of lamotrigine as an antidepressant augmentation agent in treatment-refractory unipolar depression. J Clin Psychiatry. 2011 Oct;72(10):1405-12. doi: 10.4088/JCP.09m05355gre. PMID 21367355